CLINICAL TRIAL: NCT05104307
Title: Echocardiogram and Cardiac Performance System (CPS) Ejection Fraction Validation Study
Status: Completed | Type: Observational
Sponsor: Stephen Esper (Other)
Collaborators: Sensydia Corporation (Industry)
Responsible Party: Sponsor-Investigator, Stephen Esper, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY21050167
Record Dates: First submitted 2021-10-14; First posted 2021-11-02 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Heart Diseases
Keywords: cardiovascular
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Cardiac Performance System (NSR): Subjects will wear Cardiac Performance System (CPS) non-invasive device during their standard echocardiogram
  Interventions: Device: Cardiac Performance System (CPS) Device

INTERVENTIONS:
Device: Cardiac Performance System (CPS) Device — CPS is a passive measurement system that acquires signals from multiple sensor sources that monitor cardiac heart sounds. The passive sensor systems measure sound only and do not produce energy. The CPS system also includes a Patient Monitor device that acquires data from the sensors as well as from three standard ECG electrodes. The CPS system does not acquire or store any protected health information or any subject characteristics. The CPS system has received FDA clearance K173156. Note that the CPS system was previously named Integrated CardioRespiratory (ICR) system. The CPS is FDA cleared for the ejection fraction (EF) assessment which will be its intended use for this study.

SUMMARY:
Non-significant risk device study to conduct evaluation of the performance of new device for monitoring of cardiac function (based on previous iterations 510(k) 173156)

DETAILED DESCRIPTION:
This validation study will help to establish feasibility of using the CPS monitor to screen patients for ejection fraction (EF), CO, PASP and wedge pressure compared to a standard echocardiogram. No clinical decisions will be made as a result of the CPS device EF value and this measurement will be taken for comparison purposes only.

ELIGIBILITY:
Inclusion Criteria:

• Patients over 18 scheduled for a standard echocardiogram

Exclusion Criteria:

* Patients with heart transplant history
* Patients with a Implanted Left Ventricular Assist Device (LVAD)
* Patients who have surgical scars, wounds, or bandages at the site of sensor placement
* Inadequate TTE imaging windows in left lateral position
* Otherwise deemed by the investigator as medically unfit to participate
* Chest deformities including, for example, pectus excavatum

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a standard echocardiogram
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Cardiac Performance System electronic data for Ejection Fraction | 60 minutes during Echocardiography procedure
  Cardiac function measurement including left ventricle ejection fraction to report in percentage
Cardiac Performance System electronic data for Cardiac Output | 60 minutes during Echocardiography procedure
  Cardiac function metric measurement including Cardiac Output to report in L/m
Cardiac Performance System electronic data for Pulmonary Artery Pressure | 60 minutes during Echocardiography procedure
  Cardiac function metric measurement including Pulmonary Artery Pressure to report in mmHg.
Cardiac Performance System electronic data for Pulmonary Artery Wedge Pressure | 60 minutes during Echocardiography procedure
  Cardiac function metric measurement including Pulmonary Artery Wedge Pressure to report in mmHg
Echocardiography electronic data for Ejection Fraction | 60 minutes during Echocardiography procedure
  Cardiac function measurement including left ventricle ejection fraction to report in percentage
Echocardiography electronic data for Cardiac Output | 60 minutes during Echocardiography procedure
  Cardiac function metric measurement including Cardiac Output to report in L/m
Echocardiography electronic data for Pulmonary Artery Pressure | 60 minutes during Echocardiography procedure
  Cardiac function metric measurement including Pulmonary Artery Pressure to report in mmHg.
Echocardiography electronic data for Pulmonary Artery Wedge Pressure | 60 minutes during Echocardiography procedure
  Cardiac function metric measurement including Pulmonary Artery Wedge Pressure to report in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L Esper, MD, MBA, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Montefiore Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No